CLINICAL TRIAL: NCT01308814
Title: Depression, Estrogen Replacement, and Cardiovascular Health in the Perimenopause
Brief Title: Perimenopausal Estrogen Replacement Therapy Study
Acronym: PERT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan Girdler, PhD, Principal Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-0542; R01MH087619 (NIH)
Record Dates: First submitted 2011-02-28; First posted 2011-03-04 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-07

CONDITIONS: Perimenopause; Menopause; Depression
Keywords: Perimenopause; Menopause; Depression; Cardiovascular health
MeSH Terms: conditions — Depression | interventions — Estradiol; Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo patches for 12 months and placebo pills for 12 days every 2 months.
  Interventions: Drug: Placebo
- Estradiol (Experimental): Transdermal 17β-estradiol (100 ug/day) for 12 months and oral micronized progesterone (200 mg/day) for 12 days every two months.
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — Transdermal 17β-estradiol (100 ug/day) for 12 months, administered as patches to be worn continuously and replaced once a week. Also, every 2 months, oral micronized progesterone (200 mg/day x 12 days) will be administered.
  Other Names: Climara and Prometrium.
  Arms: Estradiol
Drug: Placebo — Placebo patches for 12 months, to be worn continuously and replaced once a week. Also, placebo pills will be administered for 12 days every 2 months.
  Arms: Placebo

SUMMARY:
Study Background and Objectives: In the U.S. the majority of heart disease deaths are in women, not men. Much of the gender disparity in CVD rates relate to the burden of CV risk in women after the menopause. Depression has been associated with an increased risk for CVD morbidity and mortality. Even histories of recurrent depression in euthymic individuals are associated with elevated CV risk. Understanding the depression-CVD link may have particular relevance for women since women experience depression at a rate twice that of men. Substantial convergent evidence indicates that ovarian failure (estrogen deprivation) is one likely mechanism contributing to both CVD and depression in women. The perimenopause, a time associated with a two-fold increase in rates of depression, may provide an ideal opportunity for studying the pathophysiology of CV risk and depression in women.

The primary objective of this study is to examine the prophylactic role of estradiol in the development of depressive symptoms and the progression of cardiovascular risk in perimenopausal women with or without histories of depression. The investigators predict that women susceptible to depression will be particularly vulnerable to the acceleration of CVD in the context of the perimenopause and, consequently, will show differentially greater benefit of estradiol treatment during the menopause transition for both indices of CV risk (e.g. inflammation, endothelial function, stress reactivity), as well as depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* must be between 45 and 60 years of age
* must be in the menopause transition (irregular/ absent menstrual cycles or hot flashes)
* must be are medically healthy

Exclusion Criteria:

- currently taking antidepressant medication

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2010-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Girdler, PH.D., Principal Investigator — UNC
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Vaisar T, Gordon JL, Wimberger J, Heinecke JW, Hinderliter AL, Rubinow DR, Girdler SS, Rubinow KB. Perimenopausal transdermal estradiol replacement reduces serum HDL cholesterol efflux capacity but improves cardiovascular risk factors. J Clin Lipidol. 2021 Jan-Feb;15(1):151-161.e0. doi: 10.1016/j.jacl.2020.11.009. Epub 2020 Nov 24. PMID 33288437
- [Derived] Zannas AS, Gordon JL, Hinderliter AL, Girdler SS, Rubinow DR. IL-6 Response to Psychosocial Stress Predicts 12-month Changes in Cardiometabolic Biomarkers in Perimenopausal Women. J Clin Endocrinol Metab. 2020 Oct 1;105(10):e3757-65. doi: 10.1210/clinem/dgaa476. PMID 32706883
- [Derived] Gordon JL, Rubinow DR, Watkins L, Hinderliter AL, Caughey MC, Girdler SS. The Effect of Perimenopausal Transdermal Estradiol and Micronized Progesterone on Markers of Risk for Arterial Disease. J Clin Endocrinol Metab. 2020 May 1;105(5):e2050-60. doi: 10.1210/clinem/dgz262. PMID 31838497
- [Derived] Gordon JL, Rubinow DR, Eisenlohr-Moul TA, Xia K, Schmidt PJ, Girdler SS. Efficacy of Transdermal Estradiol and Micronized Progesterone in the Prevention of Depressive Symptoms in the Menopause Transition: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Feb 1;75(2):149-157. doi: 10.1001/jamapsychiatry.2017.3998. PMID 29322164

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Estradiol
Started | 86 | 86
Completed | 69 | 63
Not Completed | 17 | 23

BASELINE CHARACTERISTICS:
Population: Perimenopausal women.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Estradiol | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 86 | 172
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (3.0) | 50.5 (3.0) | 50.5 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 86 | 172
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 86 | 86 | 172

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms as Indicated by The Center for Epidemiologic Studies Depression Scale (CES-D)
Description: Change from pre-trial (baseline) to post-trial (month 12) in the Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D has a Range from 0-60, with higher scores indicating the presence of more symptomatology. A score of 16 or greater is indicative of clinically significant symptoms of depression.
Time Frame: Baseline, month 12
Population: The data presented here are based on individuals who completed the study and provided useable data for this particular measure at the time point reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Estradiol
Number analyzed (Participants) | 69 | 63
units on a scale | 1.04 (7.56) | -1.02 (4.89)

2. Primary Outcome: Change in Psychiatric Diagnosis as Assessed by the Structured Clinical Interview for DSM Disorders I/NP
Time Frame: Baseline and when prompted by CES-D score
Population: These data were not collected because this measure is no longer the preferred method for characterizing change in depression risk. The preferred method is now to measure depressive symptoms continuously, which was done. These continuous results can be found for the CESD score in this record.
Arm/Group | Placebo | Estradiol
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Stress Reactivity During Laboratory Session Including Trier Social Stress Test
Description: Primary measures reflecting stress reactivity will consist of mean arterial pressure (MAP), vascular resistance index (VRI), plasma cortisol, and plasma IL-6. For each of these four measures, a delta score (change from rest to stress) will be calculated and then standardized as Z scores. The individual Z scores will then be averaged to yield a single Stress Reactivity profile measure (average z score) - a composite Z score reflecting magnitude of activation in the four primary stress-responsive pathways. This composite z score at baseline will be subtracted from the composite z score at 12 months to yield this outcome measure.
Time Frame: Baseline, month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: composite Z score
Arm/Group | Placebo | Estradiol
Number analyzed (Participants) | 66 | 63
composite Z score | 0.02 (0.67) | -0.18 (0.54)

4. Secondary Outcome: Change in Functional Well-being as Assessed by the Medical Outcomes Study 36-item Short Form (SF-36)
Description: The Medical Outcomes Study 36-item Short Form (SF-36) is a measure of functional well-being, including physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to emotional health problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. The range of this scale is 0-100, where higher scores indicates a more favorable health state.
Time Frame: Baseline, month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Estradiol
Number analyzed (Participants) | 67 | 59
units on a scale | 0.94 (13.60) | 2.32 (11.32)

5. Secondary Outcome: Percentage Meeting Criteria for Metabolic Risk [Baseline and Month 12]
Description: Subjects will be classified as having metabolic risk if they either meet standard criteria for the metabolic syndrome (based on 3 of 5 risk factors: elevated blood pressure, fasting triglycerides, fasting glucose, waist circumference and low HDL-cholesterol) or they exhibit insulin resistance based on the homeostatic model assessment (HOMA) to derive HOMA-IR based on fasting insulin and glucose levels using the equation: HOMA-IR = fasting glucose (mmol/L) × fasting insulin (μU/mL)/22.5
Time Frame: Baseline, month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Estradiol
Number analyzed (Participants) | 86 | 86
Participants
  baseline with metabolic risk | 17 | 17
  12 month with metabolic risk: number analyzed (Participants) | 69 | 63
  12 month with metabolic risk | 10 | 9

6. Secondary Outcome: Change in Percentage of Brachial Artery Diameter
Description: Change (from Baseline-to-12 Month) in flow mediated dilatation (FMD) test of the brachial artery, dilatation occurs following an acute increase in blood flow, induced by via circulatory arrest in the arm for a period of time. Measured using high resolution ultrasound, yielding a measure of endothelial-dependent vasodilatation. The increase in brachial arterial diameter as a consequence of reactive hyperemia is compared to the baseline diameter of the artery and expressed as a percentage of the baseline diameter (% FMD). Flow-mediated vasodilatation at each time point was calculated as diameter of the brachial artery under reactive hyperemia minus baseline diameter of the brachial artery. The change presented here is calculated as 12 month %FMD minus baseline month %FMD.
Time Frame: Baseline, month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent flow mediated dilatation
Arm/Group | Placebo | Estradiol
Number analyzed (Participants) | 86 | 85
percent flow mediated dilatation | -0.65 (4.75) | 0.56 (4.91)

7. Secondary Outcome: Change in Baroreceptor Sensitivity
Description: A finometer noninvasive blood pressure devise (FMS) was used to collect a 10 minute recording of beat-to-beat blood pressure and pulse rate during spontaneous breathing under quiet recumbent conditions. baroreflex sensitivity was computed from the most stable 5-minute segment of this 10-minute period. Cross-spectral analysis was used to estimate the average transfer function modulus (i.e., gain) between systemic blood pressure oscillations and R-R interval oscillations in the frequency range of 0.07-0.14 Hz, also known as the low frequency band. The units of this baroreflex sensitivity (BRS) were msec/mmHg.
  The outcome presented here is the 12 month BRS minus baseline BRS.
Time Frame: Baseline, month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec/mmHg
Arm/Group | Placebo | Estradiol
Number analyzed (Participants) | 85 | 85
msec/mmHg | 0.19 (2.74) | 0.43 (2.52)

ADVERSE EVENTS:
Arm/Group | Placebo | Estradiol
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86
Other Adverse Events (participants affected / at risk) | 81/86 | 83/86
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=86) | Estradiol (N=86)
Stage 1 hypertension (Vascular disorders) | 10 | 4
High CES-D depression scale score without major or minor depression (Psychiatric disorders) | 24 | 13
Bacterial or viral infection (Infections and infestations) | 23 | 28
Bleeding changes, heavy bleeding (Blood and lymphatic system disorders) | 11 | 32
Bleeding changes, prolonged bleeding (Blood and lymphatic system disorders) | 1 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 25 | 30
Skin irritation (Skin and subcutaneous tissue disorders) | 31 | 32
Shortness of breath or chest pain (Respiratory, thoracic and mediastinal disorders) | 10 | 15
Anxiety (Psychiatric disorders) | 5 | 2
Irritability (Psychiatric disorders) | 14 | 15
Negative mood changes (Psychiatric disorders) | 25 | 20
Bleeding changes, spotting (Reproductive system and breast disorders) | 29 | 55
Bleeding changes, mild or moderate bleeding (Reproductive system and breast disorders) | 38 | 69
Bloating (Gastrointestinal disorders) | 2 | 8
Breast tenderness (Reproductive system and breast disorders) | 33 | 46
Fatigue (General disorders) | 5 | 12
GI Symptoms (Gastrointestinal disorders) | 23 | 18
Headache, not migraine (General disorders) | 58 | 52
Headache, migraine with no aura (General disorders) | 9 | 9
Hot flushes (Reproductive system and breast disorders) | 15 | 4
Leg or calf discomfort, swelling, or pain (Musculoskeletal and connective tissue disorders) | 38 | 42
Sleep issues (General disorders) | 12 | 9
Vision changes or issues (Eye disorders) | 28 | 26
Weight gain (General disorders) | 53 | 50
Other (General disorders) | 48 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No